CLINICAL TRIAL: NCT06731959
Title: A Phase 2a, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Fexlamose (AER-01) Inhalation Solution in the Treatment of Adults with Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Investigate Using Inhaled Fexlamose to Treat Adult Participants Who Have Moderate to Severe COPD
Acronym: AER-01-002
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aer Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AER-01-002
Record Dates: First submitted 2024-11-20; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fexlamose (Experimental): Fexlamose solution once daily via nebulizer for 28 days
  Interventions: Drug: Flexlamose
- Placebo (Placebo Comparator): Placebo solution once daily via nebulizer for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flexlamose — Fexlamose solution via nebulizer for 28 days
  Arms: Fexlamose
Drug: Placebo — Placebo solution via nebulizer for 28 days
  Arms: Placebo

SUMMARY:
AER-01-002 is a Phase 2a study being conducted to determine if inhaled fexlamose is an effective and safe treatment for adults with moderate to severe COPD.

Study will compare active drug to placebo.

ELIGIBILITY:
Main Inclusion Criteria

Each participant must meet all the following criteria to be enrolled in this study:

* Participant is male or female ≥40 to ≤80 years of age.
* Participant has a verified diagnosis of cigarette smoking-related COPD FEV1 that is >25% and <60% of predicted normal at Visit 1.
* Participant meets the following spirometry performance criteria:

  * Acceptability: Participant can perform acceptable spirometry (ie, meet ATS/ERS acceptability criteria) at Visits 1 and 2.
  * Repeatability: Participant can perform technically acceptable spirometry meeting repeatability criteria for FEV1 during at least 1 of the prebronchodilator assessments at Visits 1 and 2.
* Participant is on stable maintenance COPD medications with no dose adjustments for ≥4 weeks prior to Screening and during the Screening Period.
* Participant has had ≤2 COPD exacerbations requiring hospitalization in the past year.

Main Exclusion Criteria

Participants meeting any of the following criteria will be excluded from the study:

* Participant has an active uncontrolled medical condition
* Participant has a diagnosis of current asthma
* Participant has primary diagnosis of bronchiectasis, primary ciliary dyskinesia, allergic bronchopulmonary aspergillosis, or CF.
* Participant has had a COPD exacerbation in the 6 weeks prior to Visit 1
* Participant has active lung infection
* Participant has received any vaccine within 7 days prior to Day 1.
* Participant is taking a protein therapeutic for control of COPD or asthma: eg, dupilumab, tezepelumab, benralizumab, mepolizumab, omalizumab.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
FEV1 | 4 weeks
  Change from baseline in prebronchodilator FEV1 at Week 4

SECONDARY OUTCOMES:
Incidence of AEs (including SAEs and AESIs) throughout the study | 4 weeks
  Incidence of treatment related AEs (including SAEs and AESIs) throughout the study as assessed by CTCAE v4.0
Change from baseline in CT mucus plug segment score at Week 4 | 4 weeks
  Change from baseline in CT mucus plug segment score (0-20) at Week 4
Change from baseline in E-RS:COPD score at Week 4 | 4 weeks
  Change from baseline in E-RS:COPD score (0-40) at Week 4
Change from baseline in prebronchodilator FVC at Week 4 | 4 weeks
  Change from baseline in prebronchodilator forced vital capacity (FVC) at Week 4
Change from baseline in SpO2 at Week 4 | 4 weeks
  Change from baseline in oxygen saturation (SpO2) at Week 4